CLINICAL TRIAL: NCT07145034
Title: Evaluation Of Efficacy And Safety Of Prosman™ (Prunus Domestica Extract) On Prostate Function, Serum Testosterone Levels And Quality Of Life
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: All India Institute of Medical Sciences, Bhubaneswar (Other)
Responsible Party: Principal Investigator, Dr Debasish Hota, Professor, All India Institute of Medical Sciences, Bhubaneswar
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: T/IM-NF/Pharm/25-26/30
Record Dates: First submitted 2025-07-08; First posted 2025-08-28 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Healthy
Keywords: BPH

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prosman (Experimental): ProsmanTM 200 mg capsule to be taken once daily for 8 weeks
  Interventions: Drug: Prosman
- Placebo (Placebo Comparator): Placebo will be taken once daily for 8 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Prosman — Prosman, the study drug is prepared from the gummy extract (pygeum) from the Indian plum tree Prunus domestica and is available in various dosage forms. Originally, pygeum, was obtained from the African prune tree bark (Prunus africanum) and was used for the treatment of various urinary problems.
  Arms: Prosman
Other: Placebo — Placebo matched to the Prosman
  Arms: Placebo

SUMMARY:
This study is designed to test the safety and effectiveness of a plant-based supplement called Prosman™ (made from Prunus domestica extract) for men with symptoms of benign prostate hyperplasia (BPH), a common non-cancerous enlargement of the prostate gland that causes urinary problems in older men.

Key Points:

Purpose: The main goal is to see if Prosman™ can improve prostate health, hormone levels, and quality of life in men aged 40 to 60 who have BPH symptoms.

How the Study Works:

38 men will be randomly assigned to take either Prosman™ or a placebo (a dummy pill) every day for 8 weeks.

The study is randomized and controlled, meaning neither the participants nor the researchers know who is getting Prosman™ or the placebo.

Measurements:

Prostate health will be measured using a symptom score.

Blood tests will check hormone levels and other health markers.

Quality of life will also be tracked.

Safety: The study will monitor for any side effects or health problems during the trial.

Why It Matters: Current medications for BPH can have unwanted side effects, so there is interest in plant-based alternatives like Prosman™, which may offer benefits with fewer risks.

The study follows strict ethical guidelines to protect participants' privacy and safety. Data will be kept confidential, and participants can leave the study at any time.

ELIGIBILITY:
Inclusion Criteria:

* Provide voluntarily signed and dated informed consent.
* Be in good health as determined by medical history and routine blood chemistries.
* Age between 40 and 60 yr (inclusive).
* Body Mass Index of 18.5-34.9 (inclusive).
* Body weight of at least 55 kg.
* An IPSS score of 8-19 (inclusive).
* Symptoms of benign prostatic hyperplasia (BPH) for at least 6 months prior to screening (e.g. Incomplete emptying: the feeling the bladder is full, even after passing urine; Frequency: the need to pass urine often, about every one to two hours; Intermittency: the need to stop and start several times when passing urine; Urgency: feeling the urgent need to pass urine; Weak stream: a weak urine flow; Straining: trouble starting to pass urine or the need to push or strain to pass urine; Nocturia: the need to wake up at night more than two times to pass urine.
* Normotensive (seated, resting systolic blood pressure <140 mm Hg and diastolic blood pressure < 90 mm Hg. If the first measurement is slightly elevated above these limits, the subject will be given a brief (5 minute) rest period, and two more measurements will be taken. The average of all three measurements will be used to determine eligibility.
* The subject is willing and able to comply with the study protocol.

Exclusion Criteria:

* Current neurogenic bladder dysfunction.
* Current bladder neck contracture or urethral stricture.
* Current acute or chronic prostatitis or UTI.
* History of prostate cancer.
* Use of any other herbal medication for the treatment of BPH, associated symptoms, and erectile dysfunction within the past month.
* Current hematuria of unknown etiology.
* History of radiotherapy.
* History of unstable or new-onset cardiovascular/cardiorespiratory, liver, or renal conditions.
* History of diabetes or endocrine disorder.
* History of use of medications or dietary supplements known to confound the study or its endpoints.
* Alcohol consumption (more than 2 standard alcoholic drinks per day or more than 10 drinks per week) or drug abuse or dependence within the past 6 months.
* Current smokers or smoking within the past month.
* History of hyperparathyroidism or an untreated thyroid condition.
* History of malignancy in the previous 5 years except for non-melanoma skin cancer (basal cell cancer or squamous cell cancer of the skin).
* Other known gastrointestinal or metabolic conditions that might impact nutrient absorption or metabolism, e.g., short bowel syndrome, IBS/IBD, diarrheal illnesses, history of colon resection, gastro paresis, Inborn-Errors-of-Metabolism (such as PKU).
* Chronic inflammatory condition (e.g., rheumatoid arthritis, Crohn's, ulcerative colitis, Lupus, HIV/AIDS, etc.).
* Known sensitivity to any ingredient in the test formulations as listed in the product label.
* Currently participating in another research study with an investigational product or have been in another research study in the past 30 days.
* Any other conditions that, in the opinion of the medical staff, could confound the primary endpoints or place the subject at increased risk of harm if they were to participate.

Ages: 40 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The product is intended to affect prostate health
Enrollment: 38 (Estimated)
Dates: Start 2025-09-07 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Prostate health (IPSS) | 8 weeks
  To measure and compare changes in prostate health between and within groups after 8 weeks of therapy with prosmanTM The International Prostate Symptom Score (IPSS) is a questionnaire used to assess the severity of urinary symptoms in men, particularly those related to benign prostatic hyperplasia (BPH). It helps quantify the impact of these symptoms on a man's quality of life and guides treatment decisions.
  The IPSS consists of seven questions about urinary symptoms and one question about their impact on quality of life. Each symptom question is scored on a scale of 0 to 5, with higher scores indicating more severe symptoms. The quality of life question is scored from 0 to 6, with higher scores indicating a greater negative impact on quality of life.
  The total IPSS score ranges from 0 to 35.

SECONDARY OUTCOMES:
Total and free testosterone | 8 weeks
  To measure and compare changes in serum total and free testosterone between and within groups after 8 weeks of therapy
Quality of life (SF-12) | 8 weeks
  To measure and compare changes in quality of life between and within groups after 8 weeks of therapy
Glucose | 8 weeks
  To measure and compare changes in concentrations of glucose
Lipid profile | 8 weeks
  To measure and compare changes in lipid profile between and within groups.
Complete blood count | 8 weeks
  To measure and compare changes in Total and differential leucocyte count, Red blood cells count and Platelets count between and within groups.
Andogen deficiency subjective | 8 weeks
  To measure and compare changes in subjective measures of androgen deficiency by Androgen Deficiency in Aging Males questionnaire (ADAM) questionnaire.
  The ADAM questionnaire, is a screening tool used to assess potential symptoms of low testosterone in men. It's a series of yes/no questions focused on symptoms associated with androgen deficiency, such as decreased libido, fatigue, and erectile dysfunction. A positive response to the questionnaire can indicate a need for further evaluation and potential treatment for low testosterone, also known as hypogonadism between and within groups. The questionnaire typically consists of 10 questions related to symptoms like reduced libido, lack of energy, decreased strength, and erectile dysfunction.
  Scoring: A positive ADAM score is typically indicated by answering "yes" to question 1 or 7, or to at least three other questions. This suggests a potential need for further evaluation.
Electrolyte chemistry | 8 weeks
  To measure and compare changes in concentrations of calcium and electrolytes (sodium, potassium, chloride) in mMol/litre
Renal function tests -1 | 8 weeks
  To measure and compare changes in concentrations of markers of blood urea nitrogen (BUN) and creatinine in mg/dL.
Renal function tests - 2 | 8 weeks
  To measure and compare changes in concentrations of markers of total protein, and albumin IN gram/dL
Bilirubin | 8 weeks
  To measure and compare changes in concentrations of markers of liver function tests (bilirubin) in mg/dL
Liver function test | 8 weeks
  To measure and compare changes in concentrations of markers of liver function tests (alkaline phosphatase (ALP), alanine transaminase (ALT), and aspartate aminotransferase (AST)) in IU/L.
Adverse effects | 8 weeks
  To measure and compare changes in vital signs and adverse events between and within groups.

CONTACTS AND LOCATIONS:
Overall Officials: Debasish Hota, DM, Principal Investigator — AIIMS, Bhubaneswar

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Paolone DR. Benign prostatic hyperplasia. Clin Geriatr Med. 2010 May;26(2):223-39. doi: 10.1016/j.cger.2010.02.010. PMID 20497842
- [Background] Parsons JK. Modifiable risk factors for benign prostatic hyperplasia and lower urinary tract symptoms: new approaches to old problems. J Urol. 2007 Aug;178(2):395-401. doi: 10.1016/j.juro.2007.03.103. Epub 2007 Jun 11. PMID 17561143
- [Background] Thorpe A, Neal D. Benign prostatic hyperplasia. Lancet. 2003 Apr 19;361(9366):1359-67. doi: 10.1016/S0140-6736(03)13073-5. PMID 12711484
- [Background] Wilt T, Ishani A, Mac Donald R, Rutks I, Stark G. Pygeum africanum for benign prostatic hyperplasia. Cochrane Database Syst Rev. 2002;1998(1):CD001044. doi: 10.1002/14651858.CD001044. PMID 11869585
- [Background] Lees AM, Mok HY, Lees RS, McCluskey MA, Grundy SM. Plant sterols as cholesterol-lowering agents: clinical trials in patients with hypercholesterolemia and studies of sterol balance. Atherosclerosis. 1977 Nov;28(3):325-38. doi: 10.1016/0021-9150(77)90180-0. PMID 597345
- [Background] Naiyila X, Li J, Huang Y, Chen B, Zhu M, Li J, Chen Z, Yang L, Ai J, Wei Q, Liu L, Cao D. A Novel Insight into the Immune-Related Interaction of Inflammatory Cytokines in Benign Prostatic Hyperplasia. J Clin Med. 2023 Feb 24;12(5):1821. doi: 10.3390/jcm12051821. PMID 36902608